CLINICAL TRIAL: NCT00139061
Title: Phase 3 Multi-Center, Double-Blind, Randomized, Parallel Group, Forced Titration Study Of The Efficacy, Safety, And Tolerability Of Torcetrapib/Atorvastatin Compared To Fenofibrate In Subjects With Fredrickson Type IIB Dyslipidemia (Mixed Hyperlipidemia
Brief Title: Assess HDL-C Increase And Non-HDL Lowering Effect Of Torcetrapib/Atorvastatin Vs. Fenofibrate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091034
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2006-12

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — torcetrapib; Atorvastatin; Fenofibrate

INTERVENTIONS:
Drug: Torcetrapib/Atorvastatin
Drug: Fenofibrate

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To assess the HDL-C increase and non-HDL lowering effect of torcetrapib/atorvastatin vs. fenofibrate.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fredrickson Type IIB dyslipidema (Mixed Hyperlipidemia)
* Men and women at least 18 years of age

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2005-03; Study Completion 2006-05

PRIMARY OUTCOMES:
To assess HDL-C increase and non-HDL lowering effect of torcetrapib/atorvastatin vs. fenofibrate.

SECONDARY OUTCOMES:
Changes in levels of lipid parameters and other biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- France (22):
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Bordeaux Cauderan
  - Pfizer Investigational Site, Briollay
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Hagondange
  - Pfizer Investigational Site, Haut-Mauco
  - Pfizer Investigational Site, Jarny
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Mars-la-Tour
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Monguilhem
  - Pfizer Investigational Site, Mont-de-Marsan
  - Pfizer Investigational Site, Moûtiers
  - Pfizer Investigational Site, Mûrs-Erigné
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Pouilly-en-Auxois
  - Pfizer Investigational Site, Saint-Justin
  - Pfizer Investigational Site, Saint-Martin-d'Oney
  - Pfizer Investigational Site, Seysses
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Thouars
  - Pfizer Investigational Site, Tiercé